CLINICAL TRIAL: NCT04587154
Title: Womens Study to Alleviate Vasomotor Symptoms
Acronym: WAVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00045315
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Hot Flashes
Keywords: soy; menopause; hot flash
MeSH Terms: conditions — Hot Flashes | interventions — Diet, Vegan

STUDY DESIGN:
Intervention Model Description: One arm, the intervention group, has been randomly assigned to be on a low-fat vegan diet while consuming 1/2 cup of cooked soybeans each day. The other arm, the control group, will maintain their pre-study diet for the duration of the study.
Who Masked: Investigator
Masking Description: The control group will be asked to stay on their usual diet.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): This arm will follow a low-fat vegan diet in addition to 1/2 a cup of cooked soybeans each day for the duration of the study. They will also weigh themselves each week, and report weight and hot flash frequency/severity weekly.
  Interventions: Other: low-fat vegan diet with 1/2 cup soybeans daily
- Control Group (No Intervention): This arm will not change their diet for the duration of the study. They will also weigh themselves each week and report weight and hot flash frequency/severity weekly.

INTERVENTIONS:
Other: low-fat vegan diet with 1/2 cup soybeans daily — Weekly instructions will be given to the participants in the intervention group about following vegan diet with 1/2 cup of soybeans daily.
  Other Names: Vegan diet
  Arms: Intervention Group

SUMMARY:
This study tests the hypothesis that a low-fat, vegan diet including soybeans reduces the frequency and severity of menopausal hot flashes, and tests the hypothesis that total isoflavone intake is associated with the reduction in the frequency and severity of hot flashes.

DETAILED DESCRIPTION:
Women with postmenopausal hot flashes will be recruited via social media and randomly assigned to an intervention or control group. The intervention group will be asked to consume a low-fat, vegan diet including ½ cup (86g) cooked soybeans (30 g uncooked) for 12 weeks. Support will be provided by weekly meetings conducted via an Internet video conferencing platform (e.g., Zoom), along with individual counseling as needed. The control group will be asked to make no diet changes for 12 weeks but will be offered instruction in how to follow a vegan diet and about the potential role of soybeans after the 12-week point. The frequency and severity of hot flashes will be assessed before, during, and after the 12-week intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Post-menopausal women aged 40-60 years
2. English fluency
3. Moderate-to-severe hot flashes experienced at least twice per day
4. Started menopause within the last 10 years
5. No menses in preceding 12 months
6. Access to an iPhone or Android phone and willingness to install a hot-flash recording app.
7. Willingness to participate in weekly classes
8. Willingness to follow a low-fat vegan diet, including daily consumption of soybeans.

Exclusion Criteria:

1. Use of hormonal medications in the preceding 2 months
2. An explanation for hot flashes other than menopause (e.g., medication use, cancer treatment)
3. Smoking during the past six months
4. History of an eating disorder or evidence of a current eating disorder (as determined by an eating disorder diagnosis, the discretion of a qualified medical professional, or an Eating Attitudes Test-26 score >20)
5. Alcohol consumption of more than 2 drinks per day or the equivalent, episodic increased drinking (e.g., more than 2 drinks per day on weekends), or a history of alcohol abuse or dependency followed by any current use
6. Use of recreational drugs in the past 6 months
7. Use of weight-loss medications over the last 6 months or a current attempt to lose weight
8. Body Mass Index < 18.5 kg/m2
9. Soy allergy

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study only seeks people who have had their last period, thus excluding males.
Enrollment: 80 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Rate of Hot Flash | 12 weeks
  Incidents Induced by Menopause. Hot flashes will be recorded using the MyLuna application, available in the App Store for iPhone or Android.
Menopause Quality of Life Questionnaire (MENQOL) | 12 weeks
  Participants will fill out a Menopause Quality of Life Questionnaire (MENQOL)

SECONDARY OUTCOMES:
Weight Change | 12 weeks
  Body weight changes, which will be measured weekly using a Renfro scale sent out to participants in both groups.
Dietary Advanced Glycation End Products (AGEs) | 16 weeks
  Explore the effectiveness of a vegan diet in reducing dietary AGEs.
PDI, hPDI, uPDI | 16 weeks
  Assess the total plant-based index (PDI), healthy PDI, and unhealthy PDI, and their relationship with weight loss.
Ultraprocessed foods | 16 weeks
  The consumption of ultraprocessed foods will be assessed, using the NOVA classification, at baseline and 16 weeks.
Carbon Footprint | 16 weeks
  The greenhouse gas emissions (GHGE) and cumulative energy demand (CED) will be assessed, using the database of Food Impacts on the Environment for Linking to Diets (dataFIELD) and What We Eat In America (WWEIA) database, at baseline and 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Barnard, MD, FACC, Principal Investigator — President
Locations (1):
- Physicians Committee for Responsible Medicine, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American College of Obstetrics and Gynecology. Response to Women's Health Initiative Study Results by The American College of Obstetricians and Gynecologists, August 9, 2002. Internet: http://www.losolivos-obgyn.com/info/gynecology/menopause/acog_whi_2002.pdf
- [Background] Lock M. Menopause: lessons from anthropology. Psychosom Med. 1998 Jul-Aug;60(4):410-9. doi: 10.1097/00006842-199807000-00005. PMID 9710286
- [Background] Melby MK. Vasomotor symptom prevalence and language of menopause in Japan. Menopause. 2005 May-Jun;12(3):250-7. doi: 10.1097/01.gme.0000146108.27840.d9?. PMID 15879913
- [Background] Shea JL. Cross-cultural comparison of women's midlife symptom-reporting: a China study. Cult Med Psychiatry. 2006 Sep;30(3):331-62. doi: 10.1007/s11013-006-9020-4. PMID 17048096
- [Background] Melby MK, Lock M, Kaufert P. Culture and symptom reporting at menopause. Hum Reprod Update. 2005 Sep-Oct;11(5):495-512. doi: 10.1093/humupd/dmi018. Epub 2005 May 26. PMID 15919681
- [Background] Beyene Y, Martin MC. Menopausal experiences and bone density of Mayan women in Yucatan, Mexico. Am J Hum Biol. 2001 Jul-Aug;13(4):505-11. doi: 10.1002/ajhb.1082. PMID 11400221
- [Background] Nagata C, Shimizu H, Takami R, Hayashi M, Takeda N, Yasuda K. Hot flushes and other menopausal symptoms in relation to soy product intake in Japanese women. Climacteric. 1999 Mar;2(1):6-12. doi: 10.3109/13697139909025557. PMID 11910681
- [Background] Nagata C, Takatsuka N, Kawakami N, Shimizu H. Soy product intake and hot flashes in Japanese women: results from a community-based prospective study. Am J Epidemiol. 2001 Apr 15;153(8):790-3. doi: 10.1093/aje/153.8.790. PMID 11296152
- [Background] Murkies AL, Lombard C, Strauss BJ, Wilcox G, Burger HG, Morton MS. Dietary flour supplementation decreases post-menopausal hot flushes: effect of soy and wheat. Maturitas. 2008 Sep-Oct;61(1-2):27-33. doi: 10.1016/j.maturitas.2008.09.007. PMID 19434877
- [Background] Lewis JE, Nickell LA, Thompson LU, Szalai JP, Kiss A, Hilditch JR. A randomized controlled trial of the effect of dietary soy and flaxseed muffins on quality of life and hot flashes during menopause. Menopause. 2006 Jul-Aug;13(4):631-42. doi: 10.1097/01.gme.0000191882.59799.67. PMID 16837885
- [Background] Lethaby A, Marjoribanks J, Kronenberg F, Roberts H, Eden J, Brown J. Phytoestrogens for menopausal vasomotor symptoms. Cochrane Database Syst Rev. 2013 Dec 10;2013(12):CD001395. doi: 10.1002/14651858.CD001395.pub4. PMID 24323914
- [Background] Franco OH, Chowdhury R, Troup J, Voortman T, Kunutsor S, Kavousi M, Oliver-Williams C, Muka T. Use of Plant-Based Therapies and Menopausal Symptoms: A Systematic Review and Meta-analysis. JAMA. 2016 Jun 21;315(23):2554-63. doi: 10.1001/jama.2016.8012. PMID 27327802
- [Background] Thurston RC, Joffe H. Vasomotor symptoms and menopause: findings from the Study of Women's Health across the Nation. Obstet Gynecol Clin North Am. 2011 Sep;38(3):489-501. doi: 10.1016/j.ogc.2011.05.006. PMID 21961716
- [Background] Garner DM, Olmsted MP, Bohr Y, Garfinkel PE. The eating attitudes test: psychometric features and clinical correlates. Psychol Med. 1982 Nov;12(4):871-8. doi: 10.1017/s0033291700049163. PMID 6961471
- [Background] Svendsen K, Henriksen HB, Ostengen B, Jacobs DR Jr, Telle-Hansen VH, Carlsen MH, Retterstol K. Evaluation of a short Food Frequency Questionnaire to assess cardiovascular disease-related diet and lifestyle factors. Food Nutr Res. 2018 Apr 19;62. doi: 10.29219/fnr.v62.1370. eCollection 2018. PMID 29720928
- [Background] Hilditch JR, Lewis J, Peter A, van Maris B, Ross A, Franssen E, Guyatt GH, Norton PG, Dunn E. A menopause-specific quality of life questionnaire: development and psychometric properties. Maturitas. 1996 Jul;24(3):161-75. doi: 10.1016/s0378-5122(96)82006-8. PMID 8844630
- [Background] Lewis JE, Hilditch JR, Wong CJ. Further psychometric property development of the Menopause-Specific Quality of Life questionnaire and development of a modified version, MENQOL-Intervention questionnaire. Maturitas. 2005 Mar 14;50(3):209-21. doi: 10.1016/j.maturitas.2004.06.015. PMID 15734602
- [Derived] Kahleova H, Znayenko-Miller T, Holubkov R, Barnard ND. Isoflavones and changes in body weight and severe hot flashes in postmenopausal women: A secondary analysis of a randomized clinical trial. Maturitas. 2025 Sep;200:108661. doi: 10.1016/j.maturitas.2025.108661. Epub 2025 Jul 5. PMID 40663878
- [Derived] Brennan H, Znayenko-Miller T, Sutton M, Holubkov R, Barnard ND, Kahleova H. Diet quality, body weight, and postmenopausal hot flashes: a secondary analysis of a randomized clinical trial. BMC Womens Health. 2024 Nov 23;24(1):620. doi: 10.1186/s12905-024-03467-4. PMID 39580383
- [Derived] Kahleova H, Znayenko-Miller T, Uribarri J, Schmidt N, Kolipaka S, Hata E, Holtz DN, Sutton M, Holubkov R, Barnard ND. Dietary advanced glycation end-products and postmenopausal hot flashes: A post-hoc analysis of a 12-week randomized clinical trial. Maturitas. 2023 Jun;172:32-38. doi: 10.1016/j.maturitas.2023.03.008. Epub 2023 Mar 24. PMID 37084590
- [Derived] Barnard ND, Kahleova H, Holtz DN, Znayenko-Miller T, Sutton M, Holubkov R, Zhao X, Galandi S, Setchell KDR. A dietary intervention for vasomotor symptoms of menopause: a randomized, controlled trial. Menopause. 2023 Jan 1;30(1):80-87. doi: 10.1097/GME.0000000000002080. Epub 2022 Oct 16. PMID 36253903
- [Derived] Barnard ND, Kahleova H, Holtz DN, Del Aguila F, Neola M, Crosby LM, Holubkov R. The Women's Study for the Alleviation of Vasomotor Symptoms (WAVS): a randomized, controlled trial of a plant-based diet and whole soybeans for postmenopausal women. Menopause. 2021 Jul 12;28(10):1150-1156. doi: 10.1097/GME.0000000000001812. PMID 34260478